CLINICAL TRIAL: NCT00003621
Title: Phase II Trial of Pre-Irradiation Chemotherapy With BCNU, Cisplatin and Oral Etoposide Combined With Radiation Therapy in the Treatment of Grade 3 Astrocytoma (Anaplastic Astrocytoma)
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Anaplastic Astrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-987251; CDR0000066700 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Carmustine; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carmustine + etoposide + cisplatin + radiation therapy (Experimental): Patients receive carmustine IV over 1 hour on days 1-3, oral etoposide on days 1-21 and 29-49, and cisplatin IV over 1-2 hours on days 1-3 and 29-31. Treatment repeats every 8 weeks for 3 courses. Patients receive radiotherapy concurrently with the third course of chemotherapy. Quality of life is assessed every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years. Patients are followed every 3 months for 5 years and then annually thereafter.
  Interventions: Drug: carmustine; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: carmustine
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have newly diagnosed anaplastic astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of carmustine, cisplatin, and etoposide given prior to and during radiotherapy in patients with anaplastic astrocytoma. II. Assess the toxic effects associated with this regimen in these patients. III. Evaluate this regimen in terms of fatigue, depression, excessive daytime somnolence, and quality of life in these patients.

OUTLINE: Patients receive carmustine IV over 1 hour on days 1-3, oral etoposide on days 1-21 and 29-49, and cisplatin IV over 1-2 hours on days 1-3 and 29-31. Treatment repeats every 8 weeks for 3 courses. Patients receive radiotherapy concurrently with the third course of chemotherapy. Quality of life is assessed every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years. Patients are followed every 3 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, newly diagnosed, anaplastic astrocytoma No oligodendrogliomas or oligoastrocytomas

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3500/mm3 Platelet count at least 130,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 0.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled infection No concurrent malignant disease or major medical problem except superficial skin cancers

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 5 years since prior chemotherapy Endocrine therapy: Concurrent corticosteroids allowed Radiotherapy: At least 5 years since prior radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1999-02; Primary Completion 2005-02 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

SECONDARY OUTCOMES:
quality of life | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan C. Buckner, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Rao RD, Krishnan S, Fitch TR, Schomberg PJ, Dinapoli RP, Nordstrom K, Scheithauer B, O'Fallon JR, Maurer MJ, Buckner JC. Phase II trial of carmustine, cisplatin, and oral etoposide chemotherapy before radiotherapy for grade 3 astrocytoma (anaplastic astrocytoma): results of North Central Cancer Treatment Group trial 98-72-51. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):380-6. doi: 10.1016/j.ijrobp.2004.06.258. PMID 15667956
- [Result] Jaeckle K, Ballman K, O'Fallon J, et al.: Response to pre-radiation chemotherapy as a predictor of survival in patients with newly diagnosed malignant astrocytoma: a North Central Cancer Treatment Group (NCCTG) study. [Abstract] Neuro-Oncology 6 (4): TA-26, 376, 2004.